CLINICAL TRIAL: NCT01455675
Title: Phase III Study to Evaluate Clinical Efficacy and Safety of Avian Polyclonal Anti-Pseudomonas Antibodies (IgY) in Prevention of Recurrence of Pseudomonas Aeruginosa Infection in Cystic Fibrosis Patients
Brief Title: Efficacy Study of IgY (Antibody Against Pseudomonas) in Cystic Fibrosis Patients
Acronym: PsAer-IgY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mukoviszidose Institut gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PsAer-IgY
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — IgY

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IgY, gargling solution (Experimental): Avian polyclonal anti-pseudomonas antibodies (IgY), 70 ml gargling solution contains 50 mg IgY with an activity against PA, once daily
  Interventions: Drug: IgY
- Placebo, gargling solution (Placebo Comparator): 70 ml gargling solution without antibodies, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IgY — Avian polyclonal anti-pseudomonas antibodies (IgY)
  Other Names: PsAer-IgY
  Arms: IgY, gargling solution
Drug: Placebo — Placebo, 70 ml gargling solution, once daily
  Arms: Placebo, gargling solution

SUMMARY:
The purpose of this study is to prolong the time to reinfection with Pseudomonas aeruginosa after successfully treated acute or intermittent infection.

DETAILED DESCRIPTION:
This is a double -blind, placebo controlled study in which the investigational drug and the reference placebo group are gargled and swallowed. 70 ml IgY/ placebo solution is gargled every night for two minutes (for maximal 24 months) The design will include the recruitment of 144 patients randomized in two groups (72 per treatment group) In order to compensate for dropouts (i.e. patients dropping out prior to 24 months without having an event) the total sample size was planned to be approximately 180 (i.e. ~20 % dropout rate). After the actual drop-out rate has been low throughout the study, only 144 plus approx. 10% potential drop-outs were included into the study.

During the two years of treatment, subjects will be examined at the clinic every 3 months regarding safety and efficacy of the medication.

For more information please see www.impactt.eu The IMPACTT Project is funded by EU within the Framework 7 Program. PsAer-IgY Studies is part of IMPACTT Project (Workpackage 2).

ELIGIBILITY:
Inclusion Criteria:

* CF patients diagnosed according to specific clinical features and either a positive sweat chloride in double proofs or presence of disease-associated CFTR mutations in both alleles
* Males and females 5 years of age and above (being able to gargle)
* CF patients having a FEV1 value between 50% and 130% of predicted value (according to Knudson formula)
* CF patients who have had one to several sputum or throat cough swabs or endolaryngeal suction cultures positive for PA within the last three years and for whom PA has been successfully eradicated.
* Sputum / throat cough swab/ endolaryngeal suction culture negative for PA and other gram-negative bacteria on study entry.
* Patients and/ or their legal representative who are willing and able to give informed consent/ assent to participate in the study after thorough information
* Subjects of child bearing potential and who are sexually active must meet the contraception requirements (i.e. oral or injectable contraceptives, intrauterine devices, double-barrier method, contraceptive patch, male partner sterilization or condoms).

Exclusion Criteria:

* Microbiologic or serologic evidence of chronic infection with PA. Definition of chronic PA infection: Three cultures (sputum or throat cough swabs or endolaryngeal suction) have been positive for PA for 6 consecutive months (at least 3 cultures have to be taken) or more, .
* Patients, who have positive sputum culture or throat cough swab or endolaryngeal suction culture for gram-negative bacteria, such as PA, S. maltophilia, B. cepacia, A. xylosoxidans (eradication before entry in study is possible), Patients, who have positive sputum culture or throat cough swab or endolaryngeal suction culture for atypical Mycobacteria and / or Aspergillus fumigates, associated with clinical symptoms that may necessitate specific treatment.
* History of allergy/hypersensitivity to hens' egg proteins (including medication allergy) that is deemed relevant to the trial by the investigator. "Relevance" in this context refers to any increased risk of hypersensitivity reaction to trial medication.
* Patient with a known relevant substance abuse, including alcohol or drug abuse.
* Start of a new concomitant or chronic medication for CF within 4 weeks before inclusion.
* Clinically relevant diseases or medical conditions other than CF or CF-related conditions that, in the opinion of the investigator, would compromise the safety of the patient or the quality of the data. This includes, but is not limited to, significant hematological, hepatic, renal, cardiovascular, and neurological diseases (diabetic patients may participate if their disease is under good control prior to inclusion).
* Participation in another study with an investigational drug within one month or 6 half-lives (whichever is greater) preceding the inclusion.
* The patient is an employee of the investigator or the institution with direct involvement in the trial or other trials under the direction of the investigator or their members.
* Patients who are pregnant cannot be included into the study. This will be tested at inclusion visit with a urine pregnancy test (in female patients older than 10 years with secondary sexual characteristics)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-10; Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Time from start of treatment (=Day 0) to the first recurrence of PA (Pseudomonas aeruginosa) in the sputum or throat cough swab or endolaryngeal suction | max. 24 months

SECONDARY OUTCOMES:
• Change in FEV 1.0 from day 0 to each visit | max. 24 months
• Change in BMI from day 0 to each visit | max. 24 months
• Number of exacerbations | max. 24 months
• Number of days of illness in hospital and at home, i.e. out of school or work | max. 24 months
• Control of use of antibiotics, especially anti-pseudomonas antibiotics -measured as days with antibiotic treatment | max. 24 months
• Change in values of serologic tests for PA precipitins from day 0 to each visit (if applicable) | max. 24 months
• Good tolerability and comparable number and quality of adverse events like placebo group | max. 24 months
• Sputum or throat cough swab or endolaryngeal suction cultures for bacteria and fungi | max. 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Antje Schuster, Prof. Dr., Principal Investigator — University Düsseldorf
Locations (42):
- Austria (2):
  - Medizinische Universität Innsbruck Department für Kinderheilkunde, Päd III CF Zentrum, Innsbruck
  - (SALK) Universitätsklink für Kinder- und Jugendheilkunde, Ambulanz für Allergien und Lungenerkrankungen, Salzburg
- Belgium (3):
  - Clinic of Pediatric Respiratory Diseases, Infectious Diseases and Travel Clinic, Brussels
  - Hôpital Universitaire Erasme, Service de Pneumologie, Brussels
  - University Hospital Leuven, Kindergeneeskunde, Leuven
- Germany (16):
  - Charité, Christiane Herzog Zentrum, Berlin
  - Klinikum der Ruhr Universität Bochum, Bochum
  - Universitätsklinik Köln, Cologne
  - University Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Klinikum der Johann-Wolfgang- Goethe Universität Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Zentrum für Kinder- und Jugendmedizin, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - MH Hannover (adults), Hanover
  - MH Hannover (children), Hanover
  - Universitätsklinik Jena, Mukoviszidosezentrum, Jena
  - Städtisches Krankenhaus Kiel GmbH, Kiel
  - Universitätsklinikum Mainz, Mainz
  - Universitätsklinik Tübingen, Tübingen
  - Universitäts-Kinderklinik Würzburg, Würzburg
- Hungary (2):
  - Heim Pal Hospital for Children, Budapest
  - Országos Korányi TBC és Pulm. Intézet, XIX. J fsz. Kronikus-CF care, Budapest
- Ireland (4):
  - Cork University Hospital, Cork
  - Our Lady´s Children´s Hospital, Dublin
  - Tallagh Hospital, Dublin
  - Mid-Western Regional Hospital, Limerick
- Italy (4):
  - Centro Regionale Toscano di Riferimento per la Fibrosi Cistica, Florence
  - Istituto Ospedale Giannina Gaslini, Genova
  - Centro Regionale Fibrosi Cisica Lazio, Roma
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Poland (5):
  - Szpital Dzieciecy Polanki im. Macieja Plazynskiego w Gdansku sp Z o.o. Poradnia Leczenia, Gdansk
  - Centrum Medyczne Karpacz Spólka Akcyjna, Karpacz
  - Wojewódzki Szpital Specjalistyczny im. M.Kopernika Ośrodek Pediatryczny im. dr J.Korczaka, Lodz
  - NZOZ Sanatorium Cassia Villa Medica, Rabka-Zdrój
  - Instytut Matki i Dziecka Zaklad Mukowiscydozy, Warsaw
- Spain (4):
  - Hospital Universitario Cruces Neumologia, Pediatric pulmonology, Barakaldo (Vizcaya)
  - Passeig Vall d´Hebron 119, Barcelona
  - Hospital Infantil la Paz Sección de Neumologia Pediátrica, Madrid
  - Hospital Materno-Infantil Servicio de Pediatria, Málaga
- Sweden (2):
  - Karolinska University Hospital, Huddinge - CF-Centre, Stockholm
  - Uppsala University Childrens Hospital, Akademiska sjukhuset, CF center, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Information about the IMPACTT project IgY-study is part of — http://www.impactt.eu